CLINICAL TRIAL: NCT06209905
Title: Comparison of Khoury Technique Versus Titanium Reinforced PTFE Membrane in 3D Alveolar Bone Augmentation in Atrophic Posterior Mandible
Brief Title: Khoury Technique Versus Titanium Reinforced PTFE Membrane in 3D Alveolar Bone Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A06080921
Record Dates: First submitted 2024-01-06; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Alveolar Ridge Augmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ti-PTFE (Sham Comparator): A mixture of autogenous bone (scrapped from the mandibular external oblique ridge) and bovine xenograft was administered on the atrophic recipient area after decortication by low-speed reducing drills, and covered with the Ti-PTFE membrane.
  Interventions: Procedure: Alveolar ridge augmentation
- Khoury technique (Active Comparator): A bone block was harvested from the mandibular external oblique ridge, then splitted into two plates; one fixated buccally and the other fixated occlusally by bone screws), and a mixture of autogenous bone (scrapped from the mandibular external oblique ridge) and bovine xenograft was administered on the atrophic recipient area after decortication by low-speed reducing drills.
  Interventions: Procedure: Alveolar ridge augmentation

INTERVENTIONS:
Procedure: Alveolar ridge augmentation — Alveolar ridge augmentation in the three dimensions with either intervention; Ti-PTFE + bone mixture, or Khoury (Bone-plate) technique + bone mixture.

SUMMARY:
In patients with missed lower posterior teeth and resorbed lower jaw, the study aimed at restoring the jaw's height and width to accommodate placing dental implants. The study was designed as a clinical trial with two arms; control group and study group. In the control group, titanium-reinforced polytetrafluoroethylene (Ti PTFE) membrane was used to secure the grafted bone mixture in the recipient site. While in the study group, bone-plate technique (Khoury technique) for bone restoration was used to secure the grafted bone mixture as well. The donor bone was the lower jaw (for bone particles and bone-plate harvesting) and bovine bone particles mixed together to form the graft mixture. Patients were monitored for six months and assessed by X-rays. The outcome variables were volume and height of gained bone in cubic millimeters and millimeters, respectively.

DETAILED DESCRIPTION:
This study targeted bone augmentation in atrophic posterior mandible. Two groups were assigned. The first group included titanium-reinforced polytetrafluoroethylene (Ti PTFE) membrane as a rigid modality to achieve guided-bone regeneration (GBR): A mixture of autogenous bone (scrapped from the mandibular external oblique ridge) and bovine xenograft was administered on the atrophic recipient area after decortication by low-speed reducing drills, and covered with the mentioned membrane. The second group utilized rigid bone-plates (a bone block was harvested from the mandibular external oblique ridge, then splitted into two plates; one fixated buccally and the other fixated occlusally by bone screws), and the same bone mixture was prepared and introduced as in the first group. All procedures were operated under local anesthesia in a minor oral surgical setting.

Follow-up time intervals were the first postoperative day, and the sixth postoperative month. Two outcome variables were assessed; gained bone volume and gained bone height.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years old.
2. Good oral hygiene.
3. Missing mandibular posterior teeth.
4. No history of bruxism or para-functional habits.
5. Residual alveolar ridge height cannot accommodate dental implant placement.
6. Patients prepared to comply with the follow-up and maintenance program.
7. Agreement and signing the informed consent.

Exclusion Criteria:

1. Systemic diseases that may contraindicate the surgery or affect soft tissue or bone healing.
2. Heavy smoking (more than 20 cigarettes/day).
3. Intraosseous pathological lesion at the intended grafting site.
4. Gingival inflammation at the intended implant site.
5. Periodontal diseases affecting teeth adjacent to the edentulous space.
6. Inadequate inter-arch space after the indented vertical augmentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Bone volume in cubic millimeters | First postoperative day
  Volume of the gained bone was assessed by cone-beam computed tomography (CBCT)
Bone volume in cubic millimeters | Sixth postoperative month
  Volume of the gained bone was assessed by cone-beam computed tomography (CBCT)

SECONDARY OUTCOMES:
Vertical bone height in millimeters | First postoperative day
  Height of the gained bone was assessed by cone-beam computed tomography (CBCT)
Vertical bone height in millimeters | Sixth postoperative month
  Height of the gained bone was assessed by cone-beam computed tomography (CBCT)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Elkenawy, PhD, Study Director — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Addakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: No